CLINICAL TRIAL: NCT04532398
Title: Validation of the Gugging Swallowing Screen (GUSS-ICU) for the Intensive Care Unit
Brief Title: Validation of the Gugging Swallowing Screen for the Intensive Care Unit
Acronym: GUSS-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-01555; qu20Siegemund
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Dysphagia
Keywords: Gugging swallowing screen - ICU (GUSS-ICU); Gugging swallowing screen (GUSS); multi-consistency check; Flexible Endoscopic Evaluation of Swallowing (FEES)
MeSH Terms: conditions — Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Swallowing test (Other)
  Interventions: Other: Gugging swallowing screen - ICU (GUSS-ICU) index test; Other: Flexible Endoscopic Evaluation of Swallowing (FEES) reference test

INTERVENTIONS:
Other: Gugging swallowing screen - ICU (GUSS-ICU) index test — Gugging swallowing screen - ICU (GUSS-ICU) index test:
  Screening for post-extubation dysphagia: GUSS-ICU performed by 2 speech therapists independently. The GUSS-ICU model contains the core features of the original GUSS tool with the added assessment items specific to the ICU Patient (RASS score (Richmond Agitation and Sedation Scale)).
  Stage one of the screen focuses on the preliminary investigation of indirect swallowing. Stage two is comprised of varying steps that directly test swallowing. This would include the administration of semisolids, water and bread with four distinct signs that were being assessed for - deglutition, coughing, drooling and voice change. The GUSS test is evaluated using a points system (0-10) which determines the severity of dysphagia and recommends a diet form that largely minimizes the risk of aspiration. (e.g. 10 points: No dysphagia = normal food).
Other: Flexible Endoscopic Evaluation of Swallowing (FEES) reference test — Flexible Endoscopic Evaluation of Swallowing (FEES) reference test:
  Flexible Endoscopic Evaluation of Swallowing (FEES) is a technique to directly view the pharynx, larynx and esophagus during swallowing. The swallowing test is carried out first with saliva and then with different consistency (liquid, pulpy, solid) and different sized swallowing portions. This reference test is performed independently from the GUSS-ICU index test.

SUMMARY:
Aetiology of dysphagia after extubation is unknown and considered to be multifactorial. Use of a standardized dysphagia- screening permits an early diagnosis. This study is to evaluate a new GUSS (gugging swallowing Screen) tool with multi-consistency check for intensive care patients (GUSS-ICU) with dysphagia. The concurrent validity (in terms of sensitivity and specificity) of the GUSS-ICU is analyzed in comparison to the flexible endoscopic evaluation of swallowing (FEES).

DETAILED DESCRIPTION:
Aetiology of dysphagia after extubation is unknown and considered to be multifactorial. Use of a standardized dysphagia- screening permits an early diagnosis. This study is to evaluate a new GUSS (gugging swallowing Screen) tool with multi-consistency check for intensive care patients (GUSS-ICU) with dysphagia. The concurrent validity (in terms of sensitivity and specificity) of the GUSS-ICU is analyzed in comparison to the flexible endoscopic evaluation of swallowing (FEES).

The GUSS-ICU with multi-consistency check includes an indirect and a direct swallowing attempt. In indirect swallowing, the vigilance is first assessed on the basis of the RASS score (Richmond agitation-sedation scale), the presence of a stridor, the effectiveness of coughing and screeting, the possibility of swallowing saliva, drooling (saliva) and the change of voice after swallowing. If six points are reached, one can immediately proceed to the direct swallowing attempt. Unlike the original GUSS, the new GUSS-ICU direct swallowing test consists of 4 subtests with pulpy, liquid, solid and mixed solid-liquid consistency. The mixed solid-liquid consistency has been supplemented, as mixed consistencies require a more complex swallowing function with increased tongue- and lip coordination.

ELIGIBILITY:
Inclusion Criteria:

* patients treated in ICU with intubation time of at least 24 hours
* Richmond Agitation-Sedation Scale (RASS)-Score of 0 (alert and calm) to 2 (agitated)
* Inclusion in study not earlier than 1 hour after extubation
* Mini-Mental-State (MMS) Score >/=24
* signed informed consent

Exclusion Criteria:

* not capable to follow study procedures (language problems, mental disorder)
* end of life- patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity of GUSS-ICU (%) | at baseline (up to 5 hours)
  Sensitivity of GUSS-ICU for detection of dysphagia in ICU-patients after extubation (compared to FEES)
Specificity of GUSS-ICU (%) | at baseline (up to 5 hours)
  Specificity of GUSS-ICU for detection of dysphagia in ICU-patients after extubation (compared to FEES)

SECONDARY OUTCOMES:
Interrater Reliability of GUSS-ICU (Cohen's Kappa statistical analysis) | at baseline (up to 5 hours)
  Interrater Reliability of GUSS-ICU for detection of dysphagia in ICU-patients after extubation
Validity of dysphagia severity | at baseline (up to 5 hours)
  Validity of dysphagia severity (GUSS-ICU compared to FEES) by Spearman-correlation

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Troll, Principal Investigator — Logopädie (speech therapy), University Hospital Basel
Locations (1):
- Logopädie, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Troll C, Trapl-Grundschober M, Teuschl Y, Cerrito A, Compte MG, Siegemund M. A bedside swallowing screen for the identification of post-extubation dysphagia on the intensive care unit - validation of the Gugging Swallowing Screen (GUSS)-ICU. BMC Anesthesiol. 2023 Apr 13;23(1):122. doi: 10.1186/s12871-023-02072-6. PMID 37055724